CLINICAL TRIAL: NCT01125631
Title: A Phase 1, Randomized, Placebo-Controlled, Double Blind, Multicenter Study Of The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Intravenous Doses Of PF-04360365 In Japanese Patients With Mild To Moderate Alzheimer's Disease
Brief Title: Multiple Intravenous Dose Study Of PF-04360365 In Japanese Patients With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9951016
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; amyloid; antibody; Japanese
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-04360365 8.5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 8.5 mg/kg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: PF-04360365 8.5 mg/kg — 8.5 mg/kg every 8 weeks (4 doses total)
  Arms: PF-04360365 8.5 mg/kg
Drug: Placebo — Placebo every 8 weeks (4 doses total)
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the safety and tolerability of a multiple dose of PF-04360365 administered over approximately 10 minutes in Japanese patients with mild-to-moderate Alzheimer's disease and to characterize the pharmacokinetics of PF-04360365 following administration of multiple doses in Japanese patients with mild-to-moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males or females of non childbearing potential, age > or = 50
* Diagnosis of probable Alzheimer's disease, consistent with criterial from both:

  * National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
  * Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* Mini-mental status exam score of 16-26 inclusive
* Rosen-Modified Hachinski Ischemia Score of < or = 4

Exclusion Criteria:

* Diagnosis or history of other demential or neurodegenerative disorders
* Diagnosis or history of clinically significant cerebrovascular disease
* Specific findings on magnetic resonance imaging (MRI); cortical infarct, micro hemorrhage, multiple white matter lacunes, extensive white matter abnormalities
* History of autoimmune disorders
* History of allergic or anaphylactic reactions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety of PF-04360365 in Japanese subjects with mild to moderate Alzheimer's disease dosed for 6 months. (adverse events, physical/neurologic exams, vital signs, 12-lead ECG, clinical labs, brain MRI, immunogenicity and cognitive assessments) | 12 months
Pharmacokinetics of PF-04360365 following administration of multiple doses in Japanese subjects with mild to moderate Alzheimer's disease. (plasma PF-04360365 concentrations) | 12 months

SECONDARY OUTCOMES:
Plasma concentration of Aβ species following administration of multiple doses of PF-04360365 in Japanese subjects with mild to moderate Alzheimer's disease. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Pfizer Investigational Site, Hirosaki, Aomori
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Fukuyama, Hiroshima
  - Pfizer Investigational Site, Kanazawa, Ishikawa-ken

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951016&StudyName=Multiple%20Intravenous%20Dose%20Study%20Of%20PF-04360365%20In%20Japanese%20Patients%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease